CLINICAL TRIAL: NCT05256940
Title: Motivational Interviewing to Address Suicidal Ideation: A Randomized Controlled Trial With Suicidal Veterans
Brief Title: Motivational Interviewing to Address Suicidal Ideation for Veterans at High Risk for Suicide
Acronym: MI-SI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Syracuse VA Medical Center (U.S. Federal Agency); Portland VA Medical Center (U.S. Federal Agency); Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBC-001-21S; I01CX002359 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Suicide, Attempted; Suicidal Ideation
Keywords: veterans; motivational interviewing
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Motivational Interviewing to Address Suicidal Ideation (MI-SI-R) was developed to help participants at high-risk for suicide resolve their ambivalence about living by increasing their motivation to live, and is delivered in three sessions in-person, virtually, or by telephone.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment received by participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interviewing to Address Suicidal Ideation- Revised (MI-SI-R) (Experimental): Motivational Interviewing to Address Suicidal Ideation (MI-SI-R) was developed to help Veterans resolve ambivalence about living by increasing the motivation to live, and is delivered in three sessions in person, virtually, or by telephone.
  Interventions: Behavioral: Motivational Interviewing to Address Suicidal Ideation- Revised (MI-SI-R); Other: Enhanced usual care (EUC)
- Enhanced usual care (EUC) (Active Comparator): Enhanced usual care (EUC) includes safety plans administered or reviewed by research therapists, care coordination, and access to a 24-hour crisis hotline.
  Interventions: Other: Enhanced usual care (EUC)

INTERVENTIONS:
Behavioral: Motivational Interviewing to Address Suicidal Ideation- Revised (MI-SI-R) — Motivational Interviewing to Address Suicidal Ideation (MI-SI-R) was developed to help Veterans resolve ambivalence about living by increasing the motivation to live, that is delivered in three sessions in person, virtually, or by telephone.
  Arms: Motivational Interviewing to Address Suicidal Ideation- Revised (MI-SI-R)
Other: Enhanced usual care (EUC) — Enhanced usual care (EUC) includes safety plans administered or reviewed by research therapists, care coordination, and access to a 24-hour crisis hotline.

SUMMARY:
The purpose of this project is to conduct a randomized control trial with 470 Veterans to examine the impact of a revised version of Motivational Interviewing to Address Suicidal Ideation (MI-SI-R) on risk for suicide attempts and suicidal ideation when compared to high quality usual care.

DETAILED DESCRIPTION:
Research suggests that treatments to reduce suicidal behavior may need to focus on both the motivation to live and the motivation to die to obtain optimal effects. The PI developed a revised version of Motivational Interviewing to Address Suicidal Ideation (MI-SI-R) to help Veterans resolve ambivalence about living by increasing the motivation to live, that consists of three sessions delivered in-person, virtually, or by telephone. Enhanced usual care (EUC) for high-risk Veterans includes safety plans administered or reviewed by research therapists, care coordination, and access to a 24-hour crisis hotline. In a preliminary randomized controlled trial (RCT) in psychiatrically hospitalized Veterans, MI-SI-R plus EUC was associated with 50% fewer suicide attempts and 41% lower likelihood of suicidal ideation compared to EUC alone. The investigators are proposing an RCT comparing MI-SI-R plus EUC (MI-SI-R+EUC) to EUC alone in a sample of 470 high-risk Veterans with recent suicidal crises from three VHA Medical Centers, with "high-risk" defined as a suicide attempt within a month or suicidal ideation > 5 on the Beck Scale for Suicidal Ideation. Half (n = 235) will be randomized to MI-SI-R+EUC (three sessions in-person, via Video Connect, or telephone) and the remaining participants (n = 235) will receive EUC alone. All participants will be asked to complete telephone follow-up assessments at 1, 3, 6, and 12-months after randomization. This will allow the investigators to determine the efficacy of MI-SI-R+EUC in reducing risk for suicide attempts (Aim 1) and reducing overall suicidal ideation (Aim 2) when compared to EUC alone.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status,
* admitted to an inpatient unit, referred by a suicide prevention coordinator, or identified as high-risk via data extraction,
* age 18 and over,
* English speaking and reading, and
* ability to understand the study and provide informed consent,
* high-risk status confirmed by suicide attempt within a month on the Columbia- Suicide Severity Rating Scale or a score > 5 on the Scale for Suicidal Ideation

Exclusion Criteria:

* current psychosis,
* active mania,
* dementia,
* impaired decision making capacity, and
* institutionalization due to hospitalization in a non-VA facility, jail, or prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-29 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale | 12-months
  The first primary outcome is the presence (vs. absence) of non-fatal suicide attempts as reported on the Columbia-Suicide Severity Rating Scale.
Beck Scale for Suicidal Ideation | 12-month
  The second primary outcome is suicidal ideation as reported on the Beck Scale for Suicidal Ideation, which has a range from 0-38, with higher scores indicating more severe suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Britton, PhD MS, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (3):
- United States (3):
  - VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Members of the scientific community who would like a copy of limited data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing the PI at Peter.Britton@va.gov. They should state their reason for requesting the data, their plans for analyzing the data, and agree not to attempt to re-identify participants. Limited data sets will be encrypted uploaded to a protected share-point; and the password will be sent to the requestor via a separate e-mail.
Supporting Information: CSR
Time Frame: Limited data sets will be available per a Data Use Agreement (DUA), which will determine the time frame.
Access Criteria: Limited data will be provided after requestors sign a Data Use Agreement (DUA).